CLINICAL TRIAL: NCT06761794
Title: Normogram of Umbilical Artery and Fetal Middle Cerebral Artery Doppler Indices in Upper Egyptian Women
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Kamel Morsi Bakhit, Principal investigator, Assiut University
Other Study IDs: Doppler indices in normal preg
Record Dates: First submitted 2024-12-22; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Doppler in Normal Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
settle umbilical and fetal middle cerebral arteries Doppler indices( pulsatility index and resistive index) in normal pregnancy to generate a local reference range and calculate cerebroplacental ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy between 15 and 40 weeks gestational age.
2. Sure of her date (well-known LMP or confirmed date by an early ultrasound).
3. Normal fetal anatomy.
4. No history of medical disorders.

Exclusion Criteria:

1. Multiple pregnancy
2. Fetal anomalies.
3. Associated medical disorders.
4. Obstetric complications.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women with gestational age 15-40 wk, singleton fetus with no anomalies, free of medical and obstetric complications.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
pulsatility index of umbilical artery. | Through study completion, an average of 1 year
Resistive index of umbilical artery | Through study completion, an average of 1 year
pulsatility index of fetal middle cerebral artery. | Through study completion, an average of 1 year
Resistive index of fetal middle cerebral artery | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
settle cerebroplacental ratio local reference range. | Through study completion, an average of 1 year

REFERENCES:
- [Background] Acharya G, Wilsgaard T, Berntsen GK, Maltau JM, Kiserud T. Reference ranges for serial measurements of umbilical artery Doppler indices in the second half of pregnancy. Am J Obstet Gynecol. 2005 Mar;192(3):937-44. doi: 10.1016/j.ajog.2004.09.019. PMID 15746695
- [Background] Mari G. Middle cerebral artery peak systolic velocity for the diagnosis of fetal anemia: the untold story. Ultrasound Obstet Gynecol. 2005 Apr;25(4):323-30. doi: 10.1002/uog.1882. No abstract available. PMID 15789353
- [Background] Ebbing C, Rasmussen S, Kiserud T. Middle cerebral artery blood flow velocities and pulsatility index and the cerebroplacental pulsatility ratio: longitudinal reference ranges and terms for serial measurements. Ultrasound Obstet Gynecol. 2007 Sep;30(3):287-96. doi: 10.1002/uog.4088. PMID 17721916
- [Background] Maulik D, Mundy D, Heitmann E, Maulik D. Umbilical artery Doppler in the assessment of fetal growth restriction. Clin Perinatol. 2011 Mar;38(1):65-82, vi. doi: 10.1016/j.clp.2010.12.004. PMID 21353090
- [Background] Tarzamni MK, Nezami N, Gatreh-Samani F, Vahedinia S, Tarzamni M. Doppler waveform indices of fetal middle cerebral artery in normal 20 to 40 weeks pregnancies. Arch Iran Med. 2009 Jan;12(1):29-34. PMID 19111026
- [Background] Dubiel M, Breborowicz GH, Marsal K, Gudmundsson S. Fetal adrenal and middle cerebral artery Doppler velocimetry in high-risk pregnancy. Ultrasound Obstet Gynecol. 2000 Oct;16(5):414-8. doi: 10.1046/j.1469-0705.2000.00278.x. PMID 11169324